CLINICAL TRIAL: NCT00486915
Title: Concurrent Prophylactic Left Atrial Appendage Exclusion: A Randomized Controlled Trial
Brief Title: Impact of Left Atrial Appendage Exclusion on Short-Term Clinical Outcomes and Long-Term Stroke Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Dave Nagpal, Associate Professor of Cardiac Surgery and Critical Care Medicine, Surgical Director of Heart Failure and Mechanical Circulatory Support Program, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSR2007-1
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Thromboembolism; Cerebrovascular Accident
Keywords: Atrial Fibrillation; Left Atrial Appendage; Surgical Ligation; Thromboembolism; Cerebrovascular Accident
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left Atrial Appendage Exclusion (Active Comparator)
  Interventions: Procedure: Left Atrial Appendage Ligation
- Control (No Intervention)

INTERVENTIONS:
Procedure: Left Atrial Appendage Ligation
  Arms: Left Atrial Appendage Exclusion

SUMMARY:
Stroke is a major cause of morbidity in western society, and an infrequent complication of cardiac surgery. The majority of thromboembolic strokes arise from the left atrium, in particular the left atrial appendage. This study aims to assess the short-term effects of left atrial appendage ligation in terms of postoperative clinical and biochemical parameters; and the long-term effects of left atrial appendage ligation in terms of stroke incidence.

DETAILED DESCRIPTION:
In patients with non-rheumatic atrial fibrillation, the left atrial appendage is the origin of at least 90% of all left atrial clots, and the resulting systemic emboli cause approximately 25% of all strokes. The stroke rate in patients with atrial fibrillation older than 75 years of age is 8.1% per year with one clinical risk factor and is 12% per year at any age in clinical trial populations with a history of prior thromboembolism. Three-year stroke rates in elderly nursing home patients not anticoagulated are in excess of 50% (Atrial Fibrillation Investigators 1994). Anticoagulation is oftentimes withheld due to the perception of excessive risk in case of a fall; even when anticoagulation is prescribed, it is well known that therapeutic levels are not always maintained.

Left atrial appendage obliteration is commonly performed in a variety of cardiac surgical operations. There have been animal studies and theoretical arguments which demonstrate the importance of the atrial appendage in its role to support cardiac output and blood pressure, and modulate thirst and hypercoagulability (Stollberger 2003); however this has been poorly studied and documented in humans in the available literature. BNP and ANP have been shown to increase proportionately with left atrial appendage dysfunction, as have von Willebrands Factor, D-Dimer, and thrombin-antithrombin III complex (Igarashi 2001).

To date, there is not a single randomized controlled trial with adequate follow-up to assess the short- and long-term clinical effectiveness of concurrent prophylactic LAA ligation. This trial will fill that void.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mitral valve repair or replacement surgery

Exclusion Criteria:

* Patients undergoing concurrent surgical anti-arrythmia procedure
* Heart transplant patients
* Patients with known hematologic hypercoagulability disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Stroke | 4 years

SECONDARY OUTCOMES:
Short- and Long-term biochemical parameters | 1 and 5 years
Short-term clinical outcomes (Procedural complications, hospital length of stay, etc) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dave Nagpal, MD, Principal Investigator — London Health Sciences Centre; Lucia Torracca, MD, Principal Investigator — Hospital San Rafael; Ottavio Alfieri, MD, Study Director — Hospital San Rafael
Locations (1):
- Hospital San Rafael, Milan, MI, Italy